CLINICAL TRIAL: NCT03861130
Title: Genetic Determinants of Kawasaki Disease for Susceptibility and Outcome
Brief Title: Genetic Determinants of Kawasaki Disease
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Imperial College London (Other)
Collaborators: Guy's and St Thomas' NHS Foundation Trust (Other); University Hospitals Bristol and Weston NHS Foundation Trust (Other); Great Ormond Street Hospital for Children NHS Foundation Trust (Other); UK Kawasaki Support Group (Unknown); Imperial College Healthcare NHS Trust (Other); University Hospitals of North Midlands NHS Trust (Other); Burton Hospitals NHS Foundation Trust (Other); York Teaching Hospitals NHS Foundation Trust (Other); Shrewsbury and Telford Hospitals NHS Trust (Other); East Suffolk and North Essex NHS Foundation Trust (Other); New Cross Hospital (Other); Darlington Memorial Hospital (Unknown); Torbay Hospital (Unknown); Peterborough City Hospital (Unknown); University Hospitals Coventry and Warwickshire NHS Trust (Other); University Hospital of North Tees (Unknown); Cambridge University Hospitals NHS Foundation Trust (Other); Royal Cornwall Hospitals Trust (Other); Birmingham Children's Hospital (Other); University Hospital Birmingham NHS Foundation Trust (Other); Wye Valley NHS Trust (Other Government); South Tees Hospitals NHS Foundation Trust (Other); Leeds General Infirmary (Unknown); Bradford Royal Infirmary (Other); University Hospitals of Morecambe Bay NHS Trust (Other); Calderdale and Huddersfield NHS Foundation Trust (Other); St. Richard's Hospital (Other); Pinderfields General Hospital (Unknown); Worthing Hospital (Unknown); Airedale General Hospital (Unknown); Sheffield Children's NHS Foundation Trust (Other); Northwick Park Hospital (Other); West Middlesex Hospital (Unknown); Royal Albert Edward Infirmary (Unknown); Macclesfield District General Hospital (Unknown); Royal Oldham Hospital (Unknown); Stepping Hill Hospital (Unknown); North Manchester General Hospital (Unknown); Royal Bolton Hospital NHS Foundation Trust (Other); Kingston Hospital NHS Trust (Other); Tameside Hospital NHS Foundation Trust (Other); East Surrey Hospital (Unknown); St. George's Hospital, London (Other); Royal Alexandra Children's Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 13SM0678
Record Dates: First submitted 2019-03-01; First posted 2019-03-04 (Actual); Last update posted 2022-11-17 (Actual); Status verified 2022-11

CONDITIONS: Kawasaki Disease; Atypical Kawasaki Disease
Keywords: Kawasaki Disease
MeSH Terms: conditions — Mucocutaneous Lymph Node Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — EDTA, Paxgene tube, plasma, serum, urine, throat swab, saliva
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Kawasaki disease: Kawasaki disease affected children
- parent of Kawasaki disease affected child

SUMMARY:
Kawasaki disease (KD) is an acute self-limited vasculitis of infancy and early childhood. Most patients recover without sequelae although the inflammatory process causes permanent damage to the coronary arteries in 20-25% of untreated children. An infectious aetiology is suspected, but the causative agent has not been identified. The investigators aim to identify the genes underlying both susceptibility to Kawasaki disease, and the development of coronary artery aneurysms.

DETAILED DESCRIPTION:
The problem to be addressed;

Kawasaki disease is now the most common cause of acquired heart disease in children in Japan and North America. Kawasaki disease arises when genetically predisposed children encounter an as yet unidentified infectious agent which may cause only mild illness or no illness at all in children without the genetic predisposition. Other children may suffer permanent damage to the coronary arteries. Identification of the genes involved will help to improve understanding of the disease, and the development of better treatments.

Objective

The investigators aim to identify the genes underlying both susceptibility to Kawasaki disease, and the development of coronary artery aneurysms.

Design

The study will recruit nuclear families (affected child and their biological parents) through participating NHS hospitals or through the records of the UK Kawasaki Support Group.

Study size

400 affected children and both biological parents (i.e. 1200 participants)

Procedures

Informed consent using age appropriate patient/parent/guardian information sheets will be taken from parents (or from children aged 16 and over), assent will be taken from the child under the age of 16 (if appropriate). Children recruited during the acute illness; routine clinical and laboratory data and research samples (blood, urine, throat swab). Children recruited retrospectively; study questionnaire (completed by parents), saliva samples.Saliva samples from parents

ELIGIBILITY:
Inclusion Criteria:

* Affected children will be recruited if the treating clinician has made a diagnosis of possible Kawasaki disease (even if they do not fulfil the criteria below for Kawasaki disease).

The current standard diagnostic criteria for KD (Circulation 2001 103 335-336 doi: 10.1161/01.CIR 103.2.335) are:

The presence of fever for at least five days plus four of the following criteria:

1. Changes in the peripheral extremities Acute: erythema and oedema of hands and feet Convalescent: membranous desquamation of fingertips
2. Polymorphous exanthema
3. Bilateral painless bulbar conjunctival injection without exudate
4. Changes in lips and oral cavity: erythema and cracking of lips, strawberry tongue, diffuse injection of oral and pharyngeal mucosae
5. Cervical lymphadenopathy (>1.5cm diameter), usually unilateral Patients meeting not all of these criteria may meet the criteria for atypical Kawasaki disease, ie. if they have fever and two or three of the above criteria and elevation of CRP or echocardiographic evidence of coronary artery dilatation.

Parents of affected child must be biological parents.

Exclusion Criteria:

* children who do not have a diagnosis of possible Kawasaki disease

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Children under the care of consultant in hospital for Kawasaki disease, families who are members of the UK Kawasaki Support Group
Sampling Method: Probability Sample
Enrollment: 1379 (Actual)
Dates: Start 2013-02-25 (Actual); Primary Completion 2022-12-30 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Susceptibility of coronary artery aneurysms for Kawasaki patients | end date; 30 December 2022
  Identification of genes that are associated with susceptibility of coronary artery aneurysms

SECONDARY OUTCOMES:
Disease severity for Kawasaki patients | end date; 30 December 2022
  Identification of genes that are associated with disease severity

CONTACTS AND LOCATIONS:
Overall Officials: Professor M Levin, Study Chair — Imperial College London
Locations (1):
- Imperial College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No